CLINICAL TRIAL: NCT03375138
Title: A Randomized, Open-label, Parallel-group, Single-dose, Biocomparability Study of the Pharmacokinetics of Belatacept Drug Products Using Active Pharmaceutical Ingredient Manufactured by Process E PPQ Relative to Active Pharmaceutical Ingredient Manufactured by Process C in Healthy Participants
Brief Title: A Study Using Healthy Volunteers Comparing Belatacept Which Has Been Manufactured By 2 Different Processes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IM103-399
Record Dates: First submitted 2017-12-13; First posted 2017-12-15 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Healthy Volunteers
Keywords: Healthy volunteers
MeSH Terms: interventions — Abatacept

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Process E PPQ belatacept (Experimental): 10 mg/kg, single dose by intravenous (IV) infusion.
  Interventions: Drug: belatacept
- Process C belatacept (Experimental): 10 mg/kg, single dose by intravenous (IV) infusion.
  Interventions: Drug: belatacept

INTERVENTIONS:
Drug: belatacept — Specified dose on specified days

SUMMARY:
This study compares the movement of Belatacept drug products, whose active pharmaceutical ingredient has been manufactured by 2 different processes, into, through and out of the body (pharmacokinetics/PK) of healthy volunteers. Eligible participants will be randomly assigned to one of two groups, and will receive a single dose of a belatacept product once during a 4-day stay at a study site.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Healthy participants, determined by medical history, physical examination, electrocardiograms (ECGs) and clinical laboratory tests.
* Weight between 60.0 to 100.0 kg, inclusive.
* Body Mass Index (BMI) of 18.0 to 30.0 kg/m2, inclusive.
* Women of childbearing potential (WOCBP) must have a negative pregnancy test within 24 hours prior to the start of study treatment.
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment and for a total of 80 days after treatment ends.
* Women must not be breastfeeding.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment and for a total of 140 days after treatment ends. In addition, male participants must not donate sperm during this time.

Exclusion Criteria:

* Participants with active tuberculosis (TB) requiring treatment; a history of active or latent TB without documented adequate therapy; or with current clinical, radiographic or laboratory evidence fo active or latent TB.
* History of shingles (herpes zoster).
* Personal or strong family history of cancer.
* Use of tobacco- or nicotine-containing products (including, but not limited to, cigarettes, pipes, cigars, e-cigarettes, chewing tobacco, nicotine patches, nicotine lozenges, or nicotine gum) within 6 months prior to study treatment administration.
* Any known or suspected autoimmune disorder.

Other protocol defined inclusion/exclusion criteria could apply.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-05-08 (Actual); Study Completion 2019-04-02 (Actual)

PRIMARY OUTCOMES:
Area under the serum concentration-time curve from time zero extrapolated to infinite time (AUC(INF)). | Up to day 57
  Measured by plasma concentration.
Maximum observed serum concentration (Cmax). | Up to day 57
  Measured by plasma concentration.

SECONDARY OUTCOMES:
Incidence of non-serious Adverse Events (AEs). | Up to 71 days.
  Safety and tolerability as measured by incidence of non-serious AEs.
Incidence of Serious Adverse Events (SAEs). | Up to 71 days.
  Safety and tolerability as measured by incidence of SAEs.
Incidence of Adverse Events (AEs) leading to discontinuation. | Up to 71 days.
  Safety and tolerability as measured by incidence of AEs leading to discontinuation.
Number of participants with vital sign abnormalities. | Up to 71 days.
Number of participants with physical examination abnormalities. | Up to 71 days.
Number of participants with clinical laboratory abnormalities. | Up to 71 days.
Number of participants with electrocardiogram (ECG) abnormalities. | Up to 71 days.

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - PPD Austin Clinic, Austin, Texas
  - Covance, Inc., Dallas, Texas

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/Recalls/
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/pages/investigator_inquiry_form.aspx